CLINICAL TRIAL: NCT01639079
Title: Smoking Cessation Through the Web: Latino Smokers Follow-Up Study
Brief Title: Comparison of Internet Stop Smoking Intervention to Usual Care on Smoking Cessation at 6 Months
Acronym: TC5Redes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REDES-EPS-LAT-SMK-5; U01CA086117 (NIH)
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Cigarette Smoking; Nicotine Dependence
Keywords: cigarette smoking behavior; smoking cessation; Latino smoking cessation
MeSH Terms: conditions — Cigarette Smoking; Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care for Smoking (No Intervention): Usual care for smoking cessation with access to the web site after 6 months
- Internet Smoking Cessation Web Site (Experimental): Internet Stop Smoking site (TC5) offers a menu of several intervention elements from which the participants may choose as many as they wish. The links (URLs) to register for the study are:
  English: www.stopsmoking.ucsf.edu Spanish: https://www.stopsmoking.ucsf.edu/es/intro/home.aspx
  Interventions: Behavioral: Internet Smoking Cessation Web Site

INTERVENTIONS:
Behavioral: Internet Smoking Cessation Web Site — Internet Stop Smoking site (TC5) with several intervention elements from which the participants may choose as many as they wish. The links (URLs) to register for the study are: English: www.stopsmoking.ucsf.edu Spanish: https://www.stopsmoking.ucsf.edu/es/intro/home.aspx
  Other Names: Tomando Control; UCSF Stop Smoking Web Site
  Arms: Internet Smoking Cessation Web Site

SUMMARY:
The primary goal of this project is to carry out a randomized controlled trial (RCT) comparing quit rates of a Spanish/English stop smoking Web site to those of a no-intervention or "quit on your own" control. The investigators have not included a no-intervention condition in previous Web studies and although 20% of participants quit smoking at one year are 20%, obtaining evidence that the investigators interventions yield higher abstinence rates than a no-intervention control is the next logical step. Furthermore, although the investigators Web site was designed in English and Spanish, the investigators success in attracting the U.S. Hispanic/Latino (HL) population in either language has been limited, so this project only will only conduct intensive telephone follow-up of HL smokers and add new recruitment methods to do so.

DETAILED DESCRIPTION:
The main study will randomize participants to one of two conditions, an intervention condition ("immediate") and a no-intervention control ("delayed"). For the control "quit on your own" condition, we will offer a 6-month "Delayed" treatment condition (DC) and will inform participants that we are testing whether smokers who are motivated enough to seek Internet information on smoking cessation can quit on their own at the same rate as smokers who are given access to an interactive stop smoking Web site. For our intervention, the "Immediate" treatment condition (IC) is the UCSF Spanish/English Stop Smoking research Web site (www.stopsmoking.ucsf.edu) that provides smokers their preference of all elements tested in earlier trials: 1) a Web version of a National Cancer Institute-designated evidence-based intervention with updated content, the Guía para Dejar de Fumar; 2) A document summarizing pharmacological treatment to aide smoking cessation available over the counter such as nicotine gum or patch or by prescriptions from a clinician; 3) e-mail reminders to return to the site timed to individually set quit dates; 4) a mood management smoking cessation intervention; and 5) a virtual group (an asynchronous bulletin board designed to let participants provide mutual support). We will recruit study participants until we have randomized 1200 HL smokers in English or Spanish stratified by gender within language group. Participants will be followed at 1, 3, 6, and 12 months after randomization to obtain self-reported prolonged abstinence and 7- and 30-day time point prevalence rates. E-mail reminders will be sent to remind participants to return to the site to complete follow-up surveys online. Only HL smokers from the US will be followed up by telephone calls at 1 and 6 months. The main comparison measure will be cessation at 6 and 12 months from original randomization. DC participants will be able to access the interactive site after finishing the 6-month follow-up. We plan to attract Spanish-speaking HL participants to our Web site using Spanish-language TV and radio interviews and public service announcements (PSA), Spanish-language Google ads and networking with U.S. cessation groups.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* daily (smoking one or more cigarettes per day) or non-daily (smoke some days) smoker
* planning to quit within the next month
* have a valid e-mail address so to send a password required to consent online.
* speak English or Spanish
* consent to participate

Exclusion Criteria:

* does not speak English or Spanish
* age younger than 18 years
* non-smoker
* no valid email address

Note - You do not need to contact anyone to begin this study. Please access the following URLs to participate: English: www.stopsmoking.ucsf.edu Spanish: https://www.stopsmoking.ucsf.edu/es/intro/home.aspx

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2012-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
smoking abstinence | 6 months
  no cigarettes smoked in the week and/or month prior to completion of the follow-up survey

SECONDARY OUTCOMES:
Smoking fewer cigarettes | 6 months
  Reduction in the average number of cigarettes smoked per day

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo F. Muñoz, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No